CLINICAL TRIAL: NCT03135470
Title: Adequacy and Adverse Effects of Pain Medication After Ambulatory Surgery, Observational Study
Brief Title: Pain Medication After Ambulatory Surgery
Status: Terminated | Type: Observational
Why Stopped: Phase II recruitment unsuccesful, phase III lacking personnel resources
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Noora Skants, MD/PhD, Specialist in anesthesiology and intensive care, Helsinki University Central Hospital
Other Study IDs: HUS235/2017
Record Dates: First submitted 2017-04-23; First posted 2017-05-01 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Pain, Postoperative; Medication Adherence; Adverse Drug Event
Keywords: pain; ambulatory surgery; oxycodone; adverse effect
MeSH Terms: conditions — Pain, Postoperative; Medication Adherence; Drug-Related Side Effects and Adverse Reactions; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current practice group: All plenipotentiary ambulatory surgery patients, with informed consent, during the three month study period
- Standard operating protocol group: All plenipotentiary ambulatory surgery patients, with informed consent, during the three month study period after creating and informing standardized operating protocol
- Mobile phone app group: All plenipotentiary ambulatory surgery patients during the three month study period with informed consent to use mobile phone app in assesment of pain and pain medication

SUMMARY:
In Finland, there are no guidelines concerning post-operative pain medication of ambulatory surgery patients. There is a wide variety in drug prescription and medication practices of various doctors and clinics. To treat patients' pain safely, type of surgery, unique patient needs, risks, adverse effects and patient's capacity to follow instructions should be assessed during the few hour visit at the clinic. In many clinics, pain is treated after hospital discharge with strong opioid oxycodone, but the amount and dose of prescribed oxycodone varies. In Helsinki Universitys Hospital, Peijas Hospital, investigators have over 2000 ambulatory surgery procedures annually. Investigators have strict policy in oxycodone use after patient discharge compared to some other Finnish ambulatory surgery clinics. The aim of this study is to evaluate, whether the prescribed pain medication is sufficient and whether patients' suffer from adverse effects after discharge from ambulatory surgery (letter interview). The study proceeds in three phases: 1) observation of current medication practice, 2) observation after optimization and standardization of hospitals drug prescription protocol, 3) evaluation of mobile phone app in pain medication follow up.

DETAILED DESCRIPTION:
After informed consent, all patients operated as ambulatory surgery patients during the study period are given a letter interview for pain, pain medication and symptom follow up. They are also given a return envelope (with paid postal fee) to return the interview.

Based on the results of the first interview phase, our pain medication practice is reconsidered by anesthetists and surgeons to create a standard operating protocol for pain medication. The standard operating protocol is informed to personnel. Then, patient interview phase is repeated for another 3 months.

Then, investigators continue with a pilot study on using a mobile phone app in evaluating patients pain, sufficient pain medication and adverse effects. All patient with informed consent, suitable mobile phone, and willing to use it for reporting pain for hospital personnel are contacted via the mobile app. Other patients operated during that study period are interviewed by either letter interview or phone interview. Investigators try to estimate whether mobile apps are suitable for pain and medication follow-up.

ELIGIBILITY:
Inclusion Criteria:

All plenipotentiary patients, operated as ambulatory surgery patients in our clinic during the study period, with informed consent

Exclusion Criteria:

We do not accept patients, who are not plenipotentiary (minor, incompetent, prisoners, conscript in military service) or do not understand finnish or swedish written information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated as ambulatory surgery patients in our clinic (orthopaedics, urology) during 3 month study periods (three 3 month phases)
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Medication | up to two days after surgery
  all pain medication used (reported By the patient)
Pain | up to two days after surgery
  Pain assessed By the patient By numerical rating scale 0-10
Adverse effects | up to two days after surgery
  Adverse effects of the pain medication, study questions
Sufficiency of pain medication | up to two days after surgery
  Whether the pain medication used was sufficient or not, study questions

CONTACTS AND LOCATIONS:
Overall Officials: Elina Reponen, MD/PhD, Principal Investigator — Senior physician, Deputy Chief of Department
Locations (1):
- Helsinki University (Central) Hospital, Peijas Hospital, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided